CLINICAL TRIAL: NCT03644342
Title: Phase I/II Study of Niraparib With Radiotherapy for Treatment of Metastatic Invasive Carcinoma of the Cervix
Brief Title: Study of Niraparib With Radiotherapy for Treatment of Metastatic Invasive Carcinoma of the Cervix
Acronym: NIVIX
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A recent change in treatment landscape may make study futile
Sponsor: Michelle S Ludwig (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Michelle S Ludwig, Assistant Professor Radiation Oncology, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-40404
Record Dates: First submitted 2018-06-04; First posted 2018-08-23 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Carcinoma of the Cervix
Keywords: cervical cancer; Niraparib; radiotherapy; carcinoma of the cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Niraparib Arm - 100 mg (Experimental): For the purposes of this study, two dose levels of Niraparib (100 mg will be evaluated concomitant with the concurrent administration of pelvic radiotherapy.
  Interventions: Drug: Nirapaib
- Niraparib Arm - 200 mg (Experimental): For the purposes of this study, two dose levels of Niraparib (200 mg) will be evaluated concomitant with the concurrent administration of pelvic radiotherapy.
  Interventions: Drug: Nirapaib

INTERVENTIONS:
Drug: Nirapaib — (see treatment regimen and method of treatment assignment)
  Other Names: Zejula

SUMMARY:
The most effective strategy for managing distantly metastatic invasive carcinomas of the cervix is not defined. Based on the success of niraparib in breast and ovarian cancer trials and the concern for toxicities and comorbidities limiting the compliance of concurrent cisplatin for cervical cancer, this study is a phase I/II study of women diagnosed with distantly metastatic (Stage IV) disease to determine the maximum tolerated dose and to evaluate the safety, tolerability and preliminary efficacy of niraparib, an orally available small molecule PARP inhibitor when administered concurrently with definitive regional radiotherapy for treatment of cervical cancer. Women enrolled in this study will receive 3-6 cycles of induction-style carboplatin and paclitaxel followed by definitive doses of pelvic radiotherapy along with the oral niraparib given at the same time.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have histologically confirmed diagnosis of invasive squamous cell or adenocarcinoma of the cervix, FIGO Stage IIIC2 or IV (see Appendix 5 of the currently approved protocol).
2. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
3. Participant must be ≥ 18 years of age.
4. Participant must have adequate organ function within 28 days of registration, defined as follows:

   * Absolute neutrophil count ≥ 1,500/µL
   * Platelets ≥ 100,000/µL
   * Hemoglobin ≥ 9 g/dL
   * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation
   * Total bilirubin ≤ 1.5 x ULN (≤2.0 in patients with known Gilberts syndrome) OR direct bilirubin ≤ 1 x ULN
   * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
5. Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy.
6. Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
7. Female participant of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration. Pregnancy test should be repeated within 7 days before CT simulation if more than 14 days has passed since the previous pregnancy test. (If serum test is falsely positive, pregnancy can be excluded by appropriate pelvic imaging.) Patient must agree to abstain from activities that could result in pregnancy from screening through completion of 7 days of pelvic radiotherapy. Females of non-childbearing potential is defined as follows (by other than medical reasons):

   * ≥45 years of age and has not had menses for >1 year
   * Post-hysterectomy, post-bilateral oophorectomy, post external beam radiation of 6 Gy to the pelvis, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by a physical exam or imaging.
8. Participant must agree to not breastfeed during the study and for 180 days after the last dose of study treatment.
9. Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent
10. Participant must have completed 3-6 cycles of platinum based chemotherapy (acceptable regimens in Appendix 7) with clinical evidence of CR (complete response) or PR (partial response) by RECIST criteria no less than 4 weeks and no greater than 12 weeks prior to initiation of protocol therapy. If bevacizumab used, 6 weeks must elapse between administration of bevacizumab and start of radiation therapy.
11. Participant must be eligible for chemoradiation treatment in the opinion of the treating investigator.
12. Participants who are HIV+ must have CD4 counts >200/dL and demonstrate documented HAART compliance
13. Chemotherapy-related hematological toxicities must have resolved to Grade 1 or less.
14. Participant must have had a CT (chest/abdomen/pelvis) or PET-CT, within 56 days of registration

Exclusion Criteria:

1. Participant must not be simultaneously enrolled in any interventional clinical trial.
2. Participant must not have known documented intra-uterine pregnancy.
3. Participant must not have had major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.
4. Participant must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior to initiating protocol therapy. Participant that has received prior treatment with a PARP inhibitor is excluded from this study.
5. Participant last treatment with platinum based chemotherapy was ≥12 weeks from initiation of protocol therapy.
6. Participant must not receive any additional chemotherapy while on study.
7. Participant has had radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
8. Participant must not have a known hypersensitivity to niraparib components or excipients.
9. Participant must not have received colony stimulating factors (e.g. granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior to initiating protocol therapy.
10. Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
11. Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, NYHA Class III/IV heart failure, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, or any psychiatric disorder that prohibits obtaining informed consent. Participant must not have had a CVA within 6 months of registration.
12. Participant must not have had diagnosis, detection, or treatment of another type of cancer ≤ 2 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin that has been definitively treated).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle S Ludwig, MD, MPH, PhD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Luke's Medical Center McNair, Houston, Texas
  - Harris Health System - Smith Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to accrual in July 2019 and closed in September 2023 due to slow accrual and an expected change in standard care.
Pre-assignment Details: This study uses the Basian Optimal interval (BOIN)design. The initial treatment dose is 100 mg, and then for every 3 patients the dose is escalated if the observed toxicity rate at the current dose is low, de-escalated if the observed toxicity rate is high, and additional patients are treated if the observed toxicity rate is between indeterminate.
Period: Overall Study
Arm/Group | Niraparib Arm - 100 mg | Niraparib Arm - 200 mg
Started | 3 | 1 (This one patient originally was assigned on dose leve 1 (100mg) but this one patient was dosed incorrectly on dose level 2 (200mg) and was taken off-study. This patient was not evaluable for this study.)
Completed | 1 | 0
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Niraparib Arm - 100 mg | Niraparib Arm - 200 mg | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Continuous [Median (Full Range); unit: years] | 61 [41 to 66] | 40 [40 to 40] | 52 [40 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities Niraparib
Description: Maximum tolerated dose (MTD) of niraparib when administered concurrently with whole pelvic radiotherapy.
  The initial treatment dose is 100 mg, and for every 3 patients the dose is escalated and de-escalated, and additional patients are treated by the study design. Participants continue to be enrolled and assigned to treatment doses according to these rules until 17 efficacy evaluable participants are enrolled to any single dose level.
Time Frame: 7 weeks during concurrent radiation therapy and niraparib administration
Population: The study enrolled 4 patients on dose level 1(100mg). One patient was dosed incorrectly on dose leve 2 (200mg) and was taken off-study and not evaluable. There were 3 patients evaluable for this study.
Measure: Number; unit: participants
Arm/Group | Niraparib Arm - 100 mg
Number analyzed (Participants) | 3
participants
  Experienced DLT's and discontinued niraparib therapy | 2
  Tolerated niraparib at the prescribed 100mg dose without significant toxicity | 1

2. Primary Outcome: Local Progression-free Survival
Description: Local progression-free survival for patients who have received 1 or more doses of niraparib with pelvic radiation as part of their treatment for metastatic cervical cancer.
Time Frame: Up to 12 months from the time of treatment initiation to progression
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib Arm - 100 mg
Number analyzed (Participants) | 3
months | NA [NA to NA] — No patients had progression. Therefore, the median survival does not exist.

3. Secondary Outcome: Acute Toxicity Profile of Niraparib
Description: acute toxicity profile of niraparib administered concurrently with whole pelvic radiotherapy according to the CTCAE version 4 as well as the grade of each toxicity. only serious adverse events will be reported here.
Time Frame: 12 months after end of treatment, up to 1 year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Niraparib Arm - 100 mg
Number analyzed (Participants) | 3
participants | 0

4. Secondary Outcome: Quality of Life Measured Using FACT-Cx Questionnaire
Description: Functional Assessment of Cancer Therapy-Cervix (FACT Cx). It measures health related quality of life for people with cervical cancer in 4 domains: physical well being, social/family well being, emotional well being, and functional well being. All questions are a 0-4 scale. The total score is then calculated as the sum of the un-weighted subscale scores (0-27). For all FACIT scales and symptom indices, the higher the score the better the QOL
Time Frame: 12 months after end of treatment
Population: The study enrolled 4 patients on dose level 1(100mg). One patient was dosed incorrectly on dose leve 2 (200mg) and was taken off-study and not evaluable. There were 3 patients evaluable for this study. QOL data was not collected.
Arm/Group | Niraparib Arm - 100 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Tumor Response
Description: Number of tumor responses outside the radiation field using RECIST 1.1 for women receiving niraparib concurrently with whole pelvic radiotherapy. Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee (Version 1.1). Changes in only the largest unidimensional measurement (diameter) of index tumor lesions are used to assess response by RECIST criteria
Time Frame: at 28 days after completing radiation therapy (XRT completion) and at every 3 months up to 12 months
Population: as for outcome 1
Measure: Number; unit: tumors
Arm/Group | Niraparib Arm - 100 mg
Number analyzed (Participants) | 3
tumors | 0

ADVERSE EVENTS:
Time Frame: From the start of the treatment to 12 months after the end of treatment, up to 2 years.
Arm/Group | Niraparib Arm - 100 mg | Niraparib Arm - 200 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niraparib Arm - 100 mg (N=3) | Niraparib Arm - 200 mg (N=1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niraparib Arm - 100 mg (N=3) | Niraparib Arm - 200 mg (N=1)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (6) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (2)
Alkaline phosphatase increased (Investigations) | 2 (3) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 3 (15) | 1 (5)
Neutrophil count decreased (Investigations) | 2 (5) | 0 (0)
Platelet count decreased (Investigations) | 3 (11) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 3 (4) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (5) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 3 (4) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 3 (5) | 0 (0)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT03644342/Prot_SAP_000.pdf